CLINICAL TRIAL: NCT06858280
Title: Impact of Patiromer Treatment on Dietary Potassium Intake Restriction and Health-related Quality of Life and Nutrition in Patients on Chronic Dialysis Therapy: a Double-Blind, Prospective, Randomized, Placebo-Controlled, Pilot Trial
Brief Title: Patiromer and Diet/hrQoL in Chronic Dialysis
Acronym: PRINCE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRINCE; 2025-521378-33-00 (EU CTIS Number)
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Hyperkalaemia; Chronic Kidney Disease Stage 3 and 4; Dietary Intervention
MeSH Terms: conditions — Hyperkalemia; Renal Insufficiency, Chronic | interventions — patiromer

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, single-center, pilot trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patiromer (Experimental): Participants will be stratified according to the number of weekly dialysis sessions (2 vs 3) and within each stratum, and will be randomized on 1:1 basis to 3-month treatment with patiromer.
  Interventions: Drug: Patiromer 8400 MG [Veltassa]
- Placebo (Placebo Comparator): Participants will be stratified according to the number of weekly dialysis sessions (2 vs 3) and within each stratum, and will be randomized on 1:1 basis to 3-month treatment with the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Patiromer 8400 MG [Veltassa] — Randomized patients will receive one 8.4 g packet of patiromer per day or one identical packet containing a placebo. To minimize the possibility of interference with gastrointestinal absorption of other orally administered medications, administration of patiromer will be separated by at least 3 hours from other oral medicinal products. Throughout the whole study period, the study drug will be administered every day in the morning.
  Arms: Patiromer
Drug: Placebo — Randomized patients will receive one packet of placebo identical to that of patiromer. Following the same treatment sequence of patiromer, administration of the placebo will be separated by at least 3 hours from any other oral medicinal products. As for patiromer, the placebo will be administered every day in the morning.
  Arms: Placebo

SUMMARY:
This is a phase III, prospective, randomized, double-blind, placebo-controlled, single-center, pilot trial, aimed at assessing whether treatment with the oral potassium binder patiromer as compared to placebo allows withdrawal or down-titration of potassium dietary restriction without increasing the risk of hyperkalemia in chronic dialysis patients.

DETAILED DESCRIPTION:
Hyperkalemia is a major, potentially life-threatening, complication often observed in patients with end-stage kidney disease on chronic renal replacement therapy by extracorporeal hemodialysis. Restriction of dietary potassium intake is a key component of intervention strategies aimed at preventing or treating hyperkalemia and maintaining serum potassium levels in the normal range in patients on chronic dialysis therapy. However, prescription of a restrictive low-potassium diet may preclude the assumption of many potassium-rich foods such as meat, poultry, fish, milk and dairy products, fruits and vegetables and some of these foods must be boiled in water to release their potassium content, which may impact on their palatability. Thus, prescription of a diet with low potassium content may have a major impact on diet palatability and consequently on the patient's perceived quality of life. Moreover it may affect the intake of essential nutrients, such as antioxidant vitamins and fibres and alkali, with slowed intestinal transit and worsening of metabolic acidosis. Diets with restricted potassium content may result in increased sodium content and it is extremely restrictive and difficult to maintain both low potassium and low sodium intake. Finally, dialysis-dependent patients have many other dietary restrictions: they must restrict fluid (which implies not only restrictions in water and other fluids intake but also in the intake of soups and most fruits and vegetables) and sodium (which considerably affects diet palatability) intake, to prevent fluid overload and blood pressure increase with increased risk of pulmonary congestion, dyspnoea and need for additional dialysis sessions. They also must limit phosphate intake (which implies restriction of food that is particularly rich in essential nutrients such as milk and most cheeses) to prevent mineral bone disease and vascular calcifications, because phosphate is poorly cleared during the dialysis session. Finally, they also must reduce saturated fat intake because they are at increased risk of atherosclerotic disease and cardiovascular complications. Thus, potassium intake restriction is one of the several dietary restrictions that altogether have a major impact on diet palatability. Thus, the possibility to limit or avoid dietary potassium restriction would be a great relief for patients and would also have a major impact on their health status.

Historically, sodium polystyrene sulfonate (SPS) or Kayexalate® (Sanofi-Aventis S.p.A) - a resin that exchanges potassium for sodium in the large intestine - has been used as an oral potassium binder to help reduce serum potassium levels when dietary potassium restriction is not sufficient to prevent hyperkalemia or when compliance to low-potassium diet is not adequate. This medication was released into the market prior to Food and Drug Administration (FDA) creation, thus rigorous clinical trials to evaluate the risk/benefit profile of the drug are lacking, particularly in patients with Chronic Kidney Disease (CKD) and end-stage kidney disease (ESKD). SPS is a sodium-exchange resin that promotes excretion of potassium in the colon lumen with voluminous stool output and a propensity for diarrhea that is not well tolerated by most patients. In fact, in everyday clinical practice long-term SPS therapy can be associated with volume overload, hypernatremia and gastrointestinal intolerance. These side effects, in addition to the poor palatability of the resin, explain the poor compliance to the drug that is spontaneously interrupted by the majority of patients within a few weeks or months. Moreover, a Swedish observational analysis in adults with at least CKD stage IV showed that SPS treatment is associated with an excess risk of hospitalizations or death due to intestinal ischemia or thrombosis, gastrointestinal ulcers and perforation. Thus, in 2009 the FDA released a black box warning for SPS based on accumulating data showing a high incidence of colonic necrosis attributable to this compound, an event that is fatal in one-third of cases. CKD has been identified as one independent risk factor for gastrointestinal injury upon exposure to SPS. Thus, novel, safer and better-tolerated therapeutic options for the management of hyperkalemia are needed, particularly for patients with CKD.

A newer potassium binder, patiromer, has been approved by the FDA and EMA for the treatment of hyperkalemia. Patiromer is an organic, non-absorbed, sodium-free, potassium-binding polymer that exchanges potassium for calcium in the gastrointestinal tract. It has been evaluated in phase 2 and phase 3 trials showing excellent potassium-lowering efficacy, a highly predictable dose-response relationship, and a favorable side effect profile in patients with hypertension and diabetic nephropathy (AMETHYST-DN trial), heart failure with history of hyperkalemia resulting in discontinuation of RAAS inhibitors (PEARL-HF trial) or stage 3-4 CKD already treated with RAAS blockers (OPAL-HK trial). More recently, an observational outcome analysis of patients with hyperkalemia who were referred to a wide network of US dialysis centers, found that compared to a 3-month pre-index period, the occurrence and frequency of potassium baths (1K) decreased in the 3 months after initiating patiromer for hyperkalemia treatment. Consistently, 6-month patiromer treatment (8.4 g once a day or four times a week) significantly decreased serum potassium levels in 269 dialysis patients with hyperkalemia. Notably no serious adverse events have been reported with long-term use of patiromer after its introduction into the market. The most commonly reported non-serious adverse events include hypomagnesemia, diarrhea, constipation, nausea and abdominal discomfort6, events that however require treatment withdrawal in only 3% of patients. Because of the remarkably good risk/benefit profile, experts of the Kidney Disease Improving Global Outcomes (KDIGO) Controversies looking at all the available data and studies concerning potassium outcomes and treatment options, recommended including newer potassium-binding agents such as patiromer to treat hyperkalemia. Notably, patiromer compared to other potassium binders such as sodium zirconium cyclosilicate differs by exchange ion: calcium and sodium, respectively. The use of calcium rather than sodium as exchange ion may prevent the risk of sodium readsorption and secondary fluid overload that may result in excess risk of cardiovascular death and hospitalization because of heart failure in patients with or without pre-existing left ventricular dysfuction. Consistently, it is conceivable that in dialysis patients excess gastrointestinal sodium reabsorption could result in increased water intake, fluid overload and heart failure requiring fluid ultrafiltration during the dialysis session with consequent cardiovascular instability and complications. On the other hand, it is clearly demonstrated that Patiromer administered daily significantly and safely prevents hyperkalemia (with a trend to less hyperkalemia-related arrythmias) in ESKD patients on chronic dialysis therapy. The patiromer serum potassium lowering effects are confirmed by an observational, retrospective analysis showing that in 10854 patients on stable, chronic hemodialysis therapy since at least 90 days, after initiation of patiromer supplementation to prevent hyperkalemia, the percentage of patients with pre-dialysis serum potassium level < 5.5 mEq/L nearly doubled from 35.5% at baseline to 70.1% at 12 months. This increase (to 62.8%) was already apparent at two months of treatment and was observed without systematically introducing changes in diet, dialytic procedures and concomitant potassium-modifying. Another retrospective, observational, real-world study found that 3-month treatment with patiromer was associated with an average (and significant) 0.5 mEq/L decrease in serum potassium levels in 527 chronic dialysis patients referred to 2400 dialysis clinics in the United States. The results regarding dose and duration of use suggest that the providers' intention for chronic patiromer use rather than for acute or short-term potassium control18. Finally, a randomized placebo trial including also a sub-group of patients with CKD on chronic dialysis therapy showed that daily doses adjusted up to 25.2 grams according to a predefined titration algorithm (as in our present study) were safe and well tolerated over a 5-week period. No treatment-related serious adverse event was reported. Constipation and diarrhea were reported as treatment related non-serious adverse events in a few patients.

Thus, the remarkably good risk/benefit profile of patiromer in chronic hemodialysis patients provides a robust background to test in the context of a prospective, randomized controlled trial whether the potassium binding properties of patiromer can be instrumental to maintain serum potassium levels in the normal range with less restrictive (and even without) low-potassium diets and consequently improved patient-perceived quality of life. These effects are expected to translate into improved patient mental and physical health.

ELIGIBILITY:
Inclusion Criteria (to be eligible to participate in this trial, an individual must meet all the following criteria):

* More than 18-year-old
* Chronic and stable dialysis therapy with three weekly dialysis sessions for at least three months because of ESKD
* Pre-dialysis (in the long interdialytic period) serum potassium 4 to 5.5 mEq/L confirmed in two consecutive weeks, without any clinical signs or symptoms of hyperkalemia
* Stable therapy (since at least 3 months) with RAS inhibitors or MRAs. No treatment with potassium sparing diuretics
* On standardized and stable (moderately or strictly restricted) low-potassium diet
* Compliance with recommended diet
* Written informed consent

Exclusion Criteria (an individual who meets any of the following criteria will be excluded from participation in this trial):

* Hyperkalemia (pre-dialysis potassium >5.5 mEq/L during the long interdialytic period)
* Hypomagnesemia (serum magnesium <1.7 mg/dL)
* Hypercalcemia (serum calcium >10.5mg/dl)
* Ongoing treatment with potassium binding medications including Sodium polystyrene sulfonate (SPS, Kayexalate®, Sanofi-Aventis S.p.A) or Sodium zirconium cyclosilate (Lokelma®, Astra Zeneca S.p.A.)
* Ongoing treatment with potassium-sparing diuretics
* Pre-dialysis potassium <4.0 mEq/L during the long interdialytic period
* One or two weekly dialysis session
* Poor compliance to prescribed potassium-restricted diet
* History of bowel obstruction or major gastrointestinal surgery, severe gastrointestinal disorders, or swallowing disorders
* Previous history of cardiac arrhythmias potentially related to hypokalemia
* Known hypersensitivity to the active ingredient or any of the excipients of the study drug
* Inability to fully understand the potential risks and benefits related to study participation
* Concomitance of clinical conditions that could jeopardize the completion of the treatment period and/or confound data interpretation including:
* Cancer (except non-metastatic cutaneous cancers)
* Active systemic autoimmune diseases
* Concomitant treatment with steroids or any other immunosuppressive agent
* Severe/unstable heart failure requiring hospitalization or changes in pharmacological therapy or supplementary dialysis sessions over the last three months
* Refractory severe hypertension (BP >180/100 mmHg despite optimized pharmacological treatment with at least three blood pressure-lowering medications)
* Known to be positive for human immunodeficiency virus
* Drug or alcohol abuse
* Pregnancy, lactation, or intention to become pregnant before or during the study period, or within 90 days of the last dose of study treatment
* Intention to donate ova or sperm over the same period
* Childbearing potential without highly effective contraception methods according to the 2020 CTFG Recommendations related to contraception and pregnancy testing in clinical trials (https://www.hma.eu/fileadmin/dateien/Human_Medicines/01About_HMA/Working_Groups/CTFG/2020_09_HMA_CTFG_Contraception_guidance_Version_1.1_updated.pdf)
* Involvement in the study planning and/or conduct
* Participation in another clinical study with an investigational product during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Serum potassium levels | Before every dialysis session for 12 weeks after recruitment
  Change in serum potassium levels of 0.5mEq/L compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Unit, ASST Papa Giovanni XXIII, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No